CLINICAL TRIAL: NCT04974619
Title: Adaptation of an HPV Education Resource to Promote HPV Vaccination Among Latino Young Men Who Have Sex With Men in Puerto Rico and Florida -- Proyecto Hombres Previniendo el VPH (Proyecto HPV)
Brief Title: Adaptation Of An HPV Education Resource To Promote HPV Vaccination
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-20819; U54CA163068 (NIH); U54CA163071 (NIH)
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: HPV Vaccine; HPV
MeSH Terms: interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 1 Only: Online Survey group: Spanish speaking young Latino men who have sex with men (YLMSM), ages 18-26 (approximately 260 in Florida and Puerto Rico) will be asked to complete a Qualtrics survey.
  Interventions: Behavioral: Online survey
- Aim 2 Only: Interview group: Individual interviews will be conducted with key healthcare stakeholders (i.e.,healthcare clinical leadership, providers and staff, community-based organization staff)
  Interventions: Behavioral: Interviews
- Aim 3 Only: Focus Groups or Interview Group: Focus groups and/or individual interviews will be conducted in-person and/or remotely to receive feedback on the HPV vaccine education materials. Focus groups and/or individual interviews will be conducted with 24 young adult Latino men who have sex with men (YLMSM) in either English or Spanish (approximately 12 in Puerto Rico and approximately 12 in Florida). The purpose will be to gain feedback on the acceptability, accessibility, content, delivery preference, and aesthetics of the theoretically informed HPV education materials culturally targeted for Spanish- and/or English-speaking YLMSM.
  Interventions: Behavioral: Focus groups or Individual Interviews

INTERVENTIONS:
Behavioral: Online survey — Aim 1 Participants will be asked to complete a Qualtrics survey to identify knowledge gaps, health beliefs, attitudes, and educational learning preferences.
  Groups: Aim 1 Only: Online Survey group
Behavioral: Focus groups or Individual Interviews — Focus groups and/or individual interviews will be conducted in-person and/or remotely to receive feedback on the HPV vaccine education materials. Focus groups and/or individual interviews will be conducted with 24 young adult Latino men who have sex with men (YLMSM) in either English or Spanish (approximately 12 in Puerto Rico and approximately 12 in Florida). The purpose will be to gain feedback on the acceptability, accessibility, content, delivery preference, and aesthetics of the theoretically informed HPV education materials culturally targeted for Spanish- and/or English-speaking YLMSM.
  Groups: Aim 3 Only: Focus Groups or Interview Group
Behavioral: Interviews — In-depth interviews (n=20) will be conducted with key stakeholders (10 in PR and 10 in FL) eliciting feedback to inform intervention content and delivery methods and identify potential facilitators and barriers to intervention implementation.
  Groups: Aim 2 Only: Interview group

SUMMARY:
The purpose of the study is to assess Human Papillomavirus (HPV) and HPV vaccination knowledge, awareness, attitudes, health beliefs, and behaviors as well as educational preferences for learning more about HPV and HPV vaccination and to receive feedback on and adapt HPV educational materials for Young Latino Men who have Sex with Men (YLMSM).

DETAILED DESCRIPTION:
To assess HPV and HPV vaccination knowledge, awareness, attitudes, health beliefs, and behaviors as well as educational preferences among 260 Spanish-speaking YLMSM ages 18-26 in Florida and Puerto Rico. To conduct 20 in-depth interviews with key stakeholders (10 in PR and 10 in FL) eliciting feedback to inform intervention content and delivery methods and identify potential facilitators and barriers to intervention implementation. To culturally adapt an existing Cancer 101 educational resource in English and Spanish for YLMSM ages 18-26 and to conduct focus groups or individual interviews with 24 YLMSM in PR (n=12) and FL (n=12) to gain feedback on the acceptability, accessibility, content, delivery preferences, and aesthetics of the theoretically informed, HPV educational intervention targeted for English and/or Spanish-speaking YLMSM.

ELIGIBILITY:
Inclusion Criteria for Aim 1 & 3:

* Men who have had sex with a man and/or are attracted to men
* Hispanic/Latino ethnicity
* Able to read, write and understand Spanish (for Aim 1) and Spanish or English (for Aim 3)
* Aged 18-26 years
* Primary residence in either Puerto Rico or Florida
* Has access to the internet (Aim 1 only)

Additional criteria for Aim 3:

* Has regular access to a working telephone or be able to attend an in-person focus group (modifications related to COVID-19 situation will allow virtual modality to complete the focus groups or individual interviews).
* Able to read, write and understand Spanish or English

Inclusion Criteria for Aim 2:

* Individuals with a current or prior role (within last twelve months) in a community-based organization, private or public healthcare clinic, health department, college/university organization, or interest group that provides services to sexual minorities in FL or PR as a healthcare provider, staff member, group member, or in a leadership role
* Age 21 or older
* Able to understand, read and speak either Spanish or English
* Access to a working telephone or computer

Exclusion Criteria for Aim 1 & 3:

* Self identifies as either transman or transwoman
* aged <18 years or >27 years
* Individuals who contact the research team about interest in participating on Aims 1 or 3 (when recruitment cap has been completed for that aim) can be directed to Aims 1 or 3 for possible recruitment. Individuals can participate in more than 1 aim, but not more than one time in a single aim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young Latino men who have sex with men in Puerto Rico and Florida and key stakeholders (i.e., healthcare clinic leadership, providers and staff, community-based organization staff, and individuals who serve and/or have provided services to YLMSM within the past 12 months).
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Christy, PhD, Principal Investigator — Moffitt Cancer Center; Melissa Marzan-Rodriguez, DrPH, Principal Investigator — Ponce Health Sciences University
Locations (2):
- Moffitt Cancer Center, Tampa, Florida, United States
- Ponce Health Sciences University, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE

RESULTS

PARTICIPANT FLOW:
Groups:
- Aim 1 Only: Online Survey Group: Spanish speaking young Latino men who have sex with men (YLMSM), ages 18-26 (in Florida and Puerto Rico) will be asked to complete a Qualtrics survey.
  Online survey: Aim 1 Participants will be asked to complete a Qualtrics survey to identify knowledge gaps, health beliefs, attitudes, and educational learning preferences.
- Aim 2 Only: Interview Group: Individual interviews will be conducted with key healthcare stakeholders (i.e.,healthcare clinical leadership, providers and staff, community-based organization staff)
  Interviews: In-depth interviews will be conducted with key stakeholders eliciting feedback to inform intervention content and delivery methods and identify potential facilitators and barriers to intervention implementation.
- Aim 3 Only: Focus Groups or Interview Group: Each site will conduct focus groups or individual interviews with English or Spanish speaking young Latino men who have sex with men (YLMSM).
  Focus groups and/or individual interviews will be conducted in-person and/or remotely to receive feedback on the HPV vaccine education materials. Focus groups and/or individual interviews will be conducted with 24 young adult Latino men who have sex with men (YLMSM) in either English or Spanish (approximately 12 in Puerto Rico and approximately 12 in Florida). The purpose will be to gain feedback on the acceptability, accessibility, content, delivery preference, and aesthetics of the theoretically informed HPV education materials culturally targeted for Spanish- and/or English-speaking YLMSM.
Period: Overall Study
Arm/Group | Aim 1 Only: Online Survey Group | Aim 2 Only: Interview Group | Aim 3 Only: Focus Groups or Interview Group
Started | 117 | 21 (1 participant participated in Aim 2 Part 1 already. This was caught late after they were enrolled (consented and demographic data obtained). Because of their previous participation in Aim 2 Part 1, they did not complete the interview portion of Aim 2 Part 2.) | 17
Completed | 117 | 20 | 15
Not Completed | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aim 1 Only: Online Survey Group | Aim 2 Only: Interview Group | Aim 3 Only: Focus Groups or Interview Group | Total
Number analyzed (Participants) | 117 | 21 | 17 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 117 | 21 | 17 | 155
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 117 | 12 | 17 | 146
  Female | 0 | 6 | 0 | 6
  Unknown | 0 | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 117 | 11 | 17 | 145
  Not Hispanic or Latino | 0 | 6 | 0 | 6
  Unknown or Not Reported | 0 | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 26 | 2 | 0 | 28
  White | 52 | 7 | 2 | 61
  More than one race | 10 | 0 | 0 | 10
  Unknown or Not Reported | 25 | 10 | 15 | 50
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 96 | 11 | 13 | 120
  United States | 21 | 10 | 4 | 35

OUTCOME MEASURES:

1. Primary Outcome: Part 1: HPV Vaccine Knowledge (Aim 1)
Description: A scale consisting of 19 items (Score range 0-18) assessing general HPV knowledge and 9 items (Score range 0-9) assessing HPV vaccination-specific knowledge (modified from scales by Perez et al 2016 and Waller et al 2013, respectively), using a response scale consisting of True, False, and I don't know; higher scores mean higher knowledge.
Time Frame: Day 1
Population: Unvaccinated participants only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 102
score on a scale
  HPV Knowledge (Scale Score range 0-18) | 10.10 (4.87)
  HPV Vaccination Knowledge Scale (Score range 0-9) | 3.19 (2.56)

2. Primary Outcome: Part 1: HPV Vaccine Awareness (Aim 1)
Description: A scale consisting of 2 items from the Health Information National Trends Survey (HINTS) 2018, with response options Yes or No; Positive responses mean higher awareness
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 102
Participants
  Ever Heard of HPV?: No | 21
  Ever Heard of HPV?: Yes | 81
  Ever Heard of HPV Vaccine?: No | 45
  Ever Heard of HPV Vaccine?: Yes | 57

3. Primary Outcome: Part 1: HPV Vaccine Attitude (Aim 1)
Description: A scale consisting of 8 items modified from the Carolina HPV Immunization Attitudes and Beliefs Scale (CHIAS); with a 5-point response scale ranging from strongly disagree to strongly agree; higher scores mean stronger attitudes. The possible scale score range = 8-40.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 102
score on a scale | 27.38 (4.36)

4. Primary Outcome: Part 1: HPV Vaccine Health Beliefs 1 (Aim 1)
Description: Participants will complete scales; a. Perceived Risk 5 point scale from no chance to Certain I will get; higher scores mean higher perceived risk; b. Descriptive norms scale from 0% to 100%, higher score mean greater descriptive norms; c. Perceived norms 8 point scale ranging from strongly disagree to strongly agree, not applicable, higher scores mean stronger perceived norms; d. Perceived Barriers 3-point scale ranging from Not concerned at all to Very concerned, higher scores mean higher perceived barriers; e. Self-efficacy scale ranging from Strongly agree to Strongly Disagree; lower scores mean higher self-efficacy.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 102
score on a scale
  Perceived Risk. 5 point scale with of Possible scale range 5-40 | 22.81 (10.93)
  What percentage of peers do you think have received the HPV vaccine? Possible scale Range 0-100 | 20.01 (22.78)
  What percentage of male peers do you think have received HPV vaccine? Possible scale Range 0-100 | 16.26 (20.03)
  What percentage of gay/bisexual males do you think have received HPV vaccine? Possible Range 1-100 | 16.67 (19.95)
  What percentage of female peers have received the HPV vaccine? Possible Scale Range 0-100 | 24.71 (26.62)
  What percentage of gay/bisexual females received the HPV vaccine? Possible Scale Range 0-100 | 20.25 (23.02)
  Perceived Norms. 8 items. Possible Score range 8-40 | 26.55 (8.65)
  Perceived Barriers. 3 items. Possible score range 3-15. | 7.19 (3.01)
  SELFEFF1 - SELFEFF9. 9 items. Possible Score range 9-45. | 17.75 (7.05)

5. Primary Outcome: Part 1: HPV Vaccine Health Beliefs 2 (Aim 1)
Description: Count of participants who responded what they thought their perceived risk is contracting HPV. Questions range from Much below average, below average, average risk, above average risk, much above average risk, and I don't know.
Time Frame: Day 1
Population: Participants in analysis are unvaccinated.
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 102
Participants
  Much below average | 27
  Below average | 14
  Average risk (Same risk as others your age) | 29
  Above average | 6
  Much above average | 5
  I don't know | 21

6. Primary Outcome: Part 1: HPV Vaccine Health Beliefs 3 (Aim 1)
Description: Count of participants who responded within each category asking intention to get HPV vaccine among those unvaccinated, using a 7-point scale ranging from Very unlikely to Very likely, higher scores mean stronger intentions.
Time Frame: Day 1
Population: Participants in analysis are unvaccinated.
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 102
Participants
  Intention to get information about the HPV vaccine: Very Unlikey | 15
  Intention to get information about the HPV vaccine: Somewhat Unlikely | 2
  Intention to get information about the HPV vaccine: A Little Unlikely | 5
  Intention to get information about the HPV vaccine: Neither Unikely nor Likely | 13
  Intention to get information about the HPV vaccine: A Little Likely | 5
  Intention to get information about the HPV vaccine: Somewhat Likely | 26
  Intention to get information about the HPV vaccine: Very Likely | 36
  Intention to obtain more than 1 shot in the next 12 months,: Very Unlikey | 14
  Intention to obtain more than 1 shot in the next 12 months,: Somewhat Unlikely | 5
  Intention to obtain more than 1 shot in the next 12 months,: A Little Unlikely | 5
  Intention to obtain more than 1 shot in the next 12 months,: Neither Unikely nor Likely | 27
  Intention to obtain more than 1 shot in the next 12 months,: A Little Likely | 8
  Intention to obtain more than 1 shot in the next 12 months,: Somewhat Likely | 31
  Intention to obtain more than 1 shot in the next 12 months,: Very Likely | 12
  Intention to get more than one dose in the future: Very Unlikey | 12
  Intention to get more than one dose in the future: Somewhat Unlikely | 9
  Intention to get more than one dose in the future: A Little Unlikely | 4
  Intention to get more than one dose in the future: Neither Unikely nor Likely | 20
  Intention to get more than one dose in the future: A Little Likely | 2
  Intention to get more than one dose in the future: Somewhat Likely | 24
  Intention to get more than one dose in the future: Very Likely | 31

7. Primary Outcome: Part 1: HPV Vaccine Behaviors 1 (Aim 1)
Description: Count of participants who responded within each category that assesses past receipt of the HPV vaccine (modified from Brewer et al., 2009 and Brewer et al., 2017). Responses were: Yes, No, I don't know.
Time Frame: Day 1
Population: Missing data from 79 participants because orginal survey did not include this item, due to eligibility criteria at the time.
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 23
Participants
  Yes | 0
  No | 17
  I Don't Know | 6

8. Primary Outcome: Part 1: HPV Vaccine Behaviors 2 (Aim 1)
Description: Count of participants that self reported number of shots received among vaccinated individuals. Items range from 1 shot to I don't know.
Time Frame: Day 1
Population: Analysis is of vaccinated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 8
Participants
  1 Shot | 2
  2 Shots | 1
  3 Shots | 1
  At Least 1 Shot, But I Don't Know How Many | 1
  At Least 2 Shots, But I Don't Know How Many | 1
  I Don't Know | 2

9. Primary Outcome: Part 1: HPV Vaccine Educational Preferences 1 (Aim 1)
Description: A scale developed by Christy (unpublished) assessing HPV vaccine education preferences. The survey question, "Who would you like to receive information from?". Options were Physician, Other healthcare provider (Nurse, Medical Assistant), Female peer, Male peer, Parent of teen, Parent of young adult, Someone who has survived an HPV-related Cancer Other. Participants marked all that applied.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 102
Participants
  Physicians | 96
  Other Healthcare Providers | 59
  Female Peer | 8
  Male Peer | 19
  Parent of Teen | 3
  Parent of Young Adult | 4
  HPV Cancer Survivor | 40
  Other | 2

10. Primary Outcome: Part 1: HPV Vaccine Educational Preferences 2 (Aim 1)
Description: Items developed by Christy (unpublished) assessing HPV vaccine education preferences. The survey question, "Best method for delivering education?". 1 being the best method and 8 being the worst method.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 102
Participants
  In Person: 1 | 55
  In Person: 2 | 6
  In Person: 3 | 3
  In Person: 4 | 7
  In Person: 5 | 8
  In Person: 6 | 1
  In Person: 7 | 10
  In Person: 8 | 12
  Website: 1 | 13
  Website: 2 | 26
  Website: 3 | 18
  Website: 4 | 14
  Website: 5 | 9
  Website: 6 | 7
  Website: 7 | 8
  Website: 8 | 7
  Smart Phone App: 1 | 1
  Smart Phone App: 2 | 11
  Smart Phone App: 3 | 17
  Smart Phone App: 4 | 8
  Smart Phone App: 5 | 15
  Smart Phone App: 6 | 13
  Smart Phone App: 7 | 18
  Smart Phone App: 8 | 19
  Online Webinar: 1 | 2
  Online Webinar: 2 | 15
  Online Webinar: 3 | 14
  Online Webinar: 4 | 25
  Online Webinar: 5 | 15
  Online Webinar: 6 | 13
  Online Webinar: 7 | 9
  Online Webinar: 8 | 9
  Text Message: 1 | 6
  Text Message: 2 | 10
  Text Message: 3 | 13
  Text Message: 4 | 12
  Text Message: 5 | 11
  Text Message: 6 | 14
  Text Message: 7 | 19
  Text Message: 8 | 17
  Printed Booklet: 1 | 2
  Printed Booklet: 2 | 13
  Printed Booklet: 3 | 7
  Printed Booklet: 4 | 9
  Printed Booklet: 5 | 23
  Printed Booklet: 6 | 19
  Printed Booklet: 7 | 15
  Printed Booklet: 8 | 14
  Social Media Platform: 1 | 13
  Social Media Platform: 2 | 10
  Social Media Platform: 3 | 16
  Social Media Platform: 4 | 16
  Social Media Platform: 5 | 7
  Social Media Platform: 6 | 16
  Social Media Platform: 7 | 13
  Social Media Platform: 8 | 11
  Healthcare System Portal: 1 | 10
  Healthcare System Portal: 2 | 11
  Healthcare System Portal: 3 | 14
  Healthcare System Portal: 4 | 11
  Healthcare System Portal: 5 | 14
  Healthcare System Portal: 6 | 19
  Healthcare System Portal: 7 | 10
  Healthcare System Portal: 8 | 13

11. Primary Outcome: Part 1: HPV Vaccine Educational Preferences 3 (Aim 1)
Description: An item developed by Christy (unpublished) assessing HPV vaccine education preferences. The survey question, "What age would it be most helpful to for a person to receive educational information?"
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 1 Only: Online Survey Group
Number analyzed (Participants) | 102
Participants
  Ages 9-10: Missing | 89
  Ages 9-10: Check | 13
  Ages 11-14: Missing | 74
  Ages 11-14: Check | 28
  Ages 15-17: Missing | 49
  Ages 15-17: Check | 53
  Ages 18-22: Missing | 50
  Ages 18-22: Check | 52
  Ages 23-30: Missing | 70
  Ages 23-30: Check | 32
  Ages 30-45: Missing | 84
  Ages 30-45: Check | 18
  I Do Not Think So: Missing | 102
  I Do Not Think So: Check | 0

12. Primary Outcome: Part 2: Facilitators and Barriers to Intervention Implementation (Aim 2)
Description: Number of participants who consented and participated in individual interviews.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 2 Only: Interview Group
Number analyzed (Participants) | 21
Participants | 20

13. Primary Outcome: Part 3: Feedback From Focus Groups or Individual Interviews (Aim 3)
Description: Number of Participants who completed either an individual interview or participated in a focus group.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Aim 3 Only: Focus Groups/Individual Interviews: Each site will conduct focus groups or individual interviews with English or Spanish speaking young Latino men who have sex with men (YLMSM).
  Focus groups: Focus groups will be conducted in-person or remotely to evaluate the newly created educational materials about HPV vaccination. Individual interviews and/or focus groups with young Latino men who have sex with men (YLMSM) will be conducted to gain feedback on the education intervention. The purpose will be to gain feedback on the acceptability, accessibility, content, delivery preference and aesthetics of the theoretically informed, HPV education target for Spanish-speaking YLMSM.
Arm/Group | Aim 3 Only: Focus Groups/Individual Interviews
Number analyzed (Participants) | 17
Participants | 13

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected
Description: Adverse Events were not collected
Groups:
- Aim 3 Only: Focus Groups/Individual Interviews: Each site will conduct focus groups or individual interviews with English or Spanish speaking young Latino men who have sex with men (YLMSM).
  Focus groups and/or individual interviews will be conducted in-person and/or remotely to receive feedback on the HPV vaccine education materials. Focus groups and/or individual interviews will be conducted with 24 young adult Latino men who have sex with men (YLMSM) in either English or Spanish (approximately 12 in Puerto Rico and approximately 12 in Florida). The purpose will be to gain feedback on the acceptability, accessibility, content, delivery preference, and aesthetics of the theoretically informed HPV education materials culturally targeted for Spanish- and/or English-speaking YLMSM.
Arm/Group | Aim 1 Only: Online Survey Group | Aim 2 Only: Interview Group | Aim 3 Only: Focus Groups/Individual Interviews
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT04974619/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT04974619/ICF_001.pdf